CLINICAL TRIAL: NCT01669343
Title: Patient-related Predictors of Estrogen Suppression in Postmenopausal Women Using Adjuvant Letrozole
Brief Title: Aromatase Inhibitor Host Factors Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI Host Factors
Record Dates: First submitted 2012-08-15; First posted 2012-08-21 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasms
Keywords: Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-menopausal Women Using Adjuvant Letrozole (Other): Part A Routine Care Letrozole; Part B Double Dose Letrozole in overweight/obese participants
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Part A Monitor standard of care letrozole use for 28 days; measure blood levels of estrogens and vitamin D at start and end of period. Part B In overweight/obese participants who completed Part A, provide a double dose of letrozole and monitor use for 28 days; measure blood levels of estrogens and vitamin D at start and end of period.
  Other Names: Femara

SUMMARY:
The purpose of this study is to examine how key patient factors, including body size affect how well letrozole suppresses circulating estrogen levels.

This study has two components: (1) Part A - an observational phase to evaluate the impact of vitamin D and obesity on estrogen suppression in post-menopausal women already receiving letrozole treatment, and (2) Part B - an interventional phase for women with body mass index (BMI) > 25 kg/m2 to assess the effect of double AI dose on estrogen levels.

If BMI or other patient factors reduce the effectiveness of letrozole, modifications to treatment recommendations and studies to test higher dosing of letrozole may be needed to maximize the benefit of this treatment and minimize the risk of the breast cancer coming back.

DETAILED DESCRIPTION:
The available evidence suggests that circulating estradiol levels play a critical role in determining effectiveness of aromatase inhibitor therapy, and that maximal suppression of aromatase activity and estrogen production is essential for optimal disease control. Host factors such as high 25-Hydroxy Vitamin D (25-OH D) levels and obesity, which might increase residual estrogen levels, could adversely impact outcome and lead to an increased risk of recurrence or death. The primary objective of Part A (which includes women regardless of BMI) is to directly evaluate the relationship between (i) 25-OH D levels and serum estrogen levels and (ii) BMI and serum estrogen levels in a cohort of postmenopausal women on standard dose letrozole therapy (2.5 mg/day). Part B (which includes only women with BMI > 25 kg/m2) will determine whether an increased dose of letrozole (5 mg/day), which had no dose limiting side effects in a Phase I study improves suppression of estrogen in overweight/obese women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female patients
* histological confirmed diagnosis of estrogen receptor and/or progesterone receptor positive breast cancer (Stage I-III) who have completed local therapy
* Currently prescribed and taking letrozole 2.5 mg daily for a minimum of 3 months
* Willing to provide written informed consent to participate
* for the experimental arm: all of the above and body mass index (BMI) > 25 kg/m2

Exclusion Criteria:

* Known abnormal liver or renal function defined by:

  1. Serum Creatinine > 1.25 times institutional upper limit of normal (ULN) or Calculated Creatinine Clearance < 40 mL/min
  2. Serum Bilirubin, Aspartate transaminase (AST) or alanine transaminase (ALT) > 1.5 times ULN
* Presence of persistent local or known metastatic cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, M.D., Principal Investigator — Princess Margaret Hospital, Canada
Locations (3):
- Canada (3):
  - Princess Margaret Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the related manuscript are kept in institutional file storage on an internal server at Lunenfeld-Tanenbaum Research Institute. There are de-identification concerns in small, regionally restricted, clinical datasets which prevent these data being openly available, but data will be made available at reasonable request from the corresponding author for up to and including 5 years from publication of the related manuscript.
  For all data requests please contact:
  Dr David Cescon, Princess Margaret Cancer Centre, University Health Network, Toronto, Ontario, Canada. Dave.Cescon@uhn.ca
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Up to and including 5 years from publication of the related manuscript (Elliott, Mitchell J et al. "Association between BMI, vitamin D, and estrogen levels in postmenopausal women using adjuvant letrozole: a prospective study." NPJ breast cancer vol. 6 22. 12 Jun. 2020)
Access Criteria: Reasonable request

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-menopausal Women Using Adjuvant Letrozole: Part A: All patients enrolled, on standard of care letrozole; Part B: All patients with BMI>=25 who completed Part A, on a double dose of letrozole
Period: Part A: All Patients
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Started | 121
Completed | 112
Not Completed | 9
Not completed — Withdrawal by Subject | 7
Not completed — Ineligibility discovered after enrollment | 2
Period: Part B: Patients With BMI>=25
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Started (By study design, only patients with BMI>=25 was eligible for Part B) | 48
Completed | 31
Not Completed | 17
Not completed — Withdrawal by Subject | 13
Not completed — Recruited during interim analysis | 3
Not completed — Ineligibility discovered after enrollment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 112
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only overweight/obese participant who completed Part A were enrolled in Part B
  years
    Part A | 61.7 (7.6)
    Part B: number analyzed (Participants) | 31
    Part B | 61.0 (66)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only overweight/obese participant who completed Part A were enrolled in Part B
  Participants
    Part A: Female | 112
    Part A: Male | 0
    Part B: number analyzed (Participants) | 31
    Part B: Female | 31
    Part B: Male | 0
Age at menopause [Mean (Standard Deviation); unit: years] — Population: Only overweight/obese participant who completed Part A were enrolled in Part B
  years
    Part A | 49.2 (4.7)
    Part B: number analyzed (Participants) | 31
    Part B | 48.4 (5.2)
Vitamin D supplementation [Count of Participants; unit: Participants] — Population: Only overweight/obese participant who completed Part A were enrolled in Part B
  Participants
    Part A | 109
    Part B: number analyzed (Participants) | 31
    Part B | 31
Letrozole use prior to study [Mean (Standard Deviation); unit: months] | 18.1 (17.6)

OUTCOME MEASURES:

1. Primary Outcome: Part A Correlation of Day 29 Estradiol With BMI
Description: Determine if estradiol levels vary with BMI levels after 28 days of monitored adherence to standard dose letrozole, by calculating the Pearson correlation between estradiol and log-transformed BMI
Time Frame: Day 29
Population: Part A
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 112
correlation coefficient | 0.06 [-0.13 to 0.24]

2. Primary Outcome: Part A Correlation of Day 29 Estrone With BMI
Description: Determine if estrone levels vary with BMI levels after 28 days of monitored adherence to standard dose letrozole, by calculating the Pearson correlation between estrone and log-transformed BMI
Time Frame: Day 29
Population: Part A
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 112
correlation coefficient | 0.07 [-0.12 to 0.25]

3. Primary Outcome: Part A Correlation of Day 29 Estradiol With Vitamin D
Description: Determine if estradiol levels vary with Vitamin D levels levels after 28 days of monitored adherence to standard dose letrozole, by calculating the Pearson correlation between estradiol and log-transformed Vitamin D level
Time Frame: Day 29
Population: Part A
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 112
correlation coefficient | -0.04 [-0.22 to 0.15]

4. Primary Outcome: Part A Correlation of Day 29 Estrone With Vitamin D
Description: Determine if estrone levels vary with Vitamin D levels levels after 28 days of monitored adherence to standard dose letrozole, by calculating the Pearson correlation between estrone and log-transformed Vitamin D level
Time Frame: Day 29
Population: Part A
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 112
correlation coefficient | 0.04 [-0.14 to 0.23]

5. Primary Outcome: Part B Change in Estradiol Level After Double Dose of Letrozole
Description: In overweight/obese patients enrolled in part B, determine if blood levels of estradiol levels changed from before to after the double dose of letrozole
Time Frame: Day 29 to Day 58
Population: Part B participants
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 31
pmol/L | 0.1 [-0.56 to 0.78]

6. Secondary Outcome: Plasma Letrozole
Time Frame: Day 29 and day 58
Population: Data were not collected
Groups:
- Post-menopausal Women Using Adjuvant Letrozole: Part B Double Dose Letrozole in overweight/obese participants
  Part B: In overweight/obese participants who completed Part A, provide a double dose of letrozole and monitor use for 28 days; measure blood levels of estrogens and vitamin D at start and end of period.
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 0

7. Secondary Outcome: Endocrine Symptoms During Part A of Study
Description: Functional Assessment of Cancer Therapy - Endocrine Sub-scale (FACT-ES) consists of 19 questions answered of a Likert scale. The sub-scale score ranges from 0 to 76 and the higher the score the better the quality of life
Time Frame: baseline, day 29 (end of part A)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Post-menopausal Women Using Adjuvant Letrozole: Part A: All patients enrolled, on standard of care letrozole
Arm/Group | Post-menopausal Women Using Adjuvant Letrozole
Number analyzed (Participants) | 112
score on a scale
  Day 1 | 62.4 (9.6)
  Day 29 | 62.9 (10.4)

8. Other Pre Specified Outcome: Musculoskeletal Symptoms
Time Frame: baseline (day 1), day 29 (end of part A) and day 58 (end of part B)
Reporting Status: Not Posted

9. Secondary Outcome: Endocrine Symptoms During Part B of the Study
Description: as for outcome 7
Time Frame: day 29 (end of part A) and day 58 (end of part B)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part B: Part B: Patients With BMI>=25, on double dose of letrozole
Arm/Group | Part B
Number analyzed (Participants) | 31
score on a scale
  Day 29 | 61.7 (11.1)
  Day 58 | 61.2 (11.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of the study: 29 days for patients taking part in Part A only, 58 days for patients that took part in Parts A and B
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.01
Groups:
- Full Study: Adverse events collected during part A, 29 days of monitored adherence to standard of care letrozole and Part B .
Arm/Group | Full Study
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 2/121
Other Adverse Events (participants affected / at risk) | 8/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Study (N=121)
Renal Colic/Constipation (Renal and urinary disorders) | 1 (1) — Hospitalized for grade 3 Renal Colic/Constipation
Stroke (Vascular disorders) | 1 (1) — Hospitalized for stroke, grade 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Study (N=121)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No